CLINICAL TRIAL: NCT07353398
Title: Early-phase Clinical Study on Safety, Tolerability and Preliminary Efficacy of ART002g1 Injection in the Treatment of Heterozygous Familial Hypercholesterolemia
Brief Title: Early-phase Study of ART002g1 Injection in HeFH: Safety, Tolerability and Preliminary Efficacy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Accuredit Therapeutics US Limited (Industry)
Responsible Party: Principal Investigator, Rong Jiang, Associate Chief Physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-ATMP-2026001
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Heterozygous Familial Hypercholesterolemia
Keywords: ART002g1; LNP; HeFH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: ART002g1 Injection - Dose Group 1 ( Single IV Infusion) (Experimental): Participants will receive a single dose of ART002g1.
  Interventions: Drug: ART002g1 Injection
- Experimental: ART002g1 Injection - Dose Group 2 (Single IV Infusion) (Experimental): Participants will receive a single dose of ART002g1.
  Interventions: Drug: ART002g1 Injection
- Experimental: ART002g1 Injection - Extended Dose Group ( Single IV Infusion) (Experimental): Participants will receive a single Optimal Biological Dose (OBD) of ART002g1, which is based on the results of the ascending dose escalation.
  Interventions: Drug: ART002g1 Injection

INTERVENTIONS:
Drug: ART002g1 Injection — Intravenous (IV) infusion

SUMMARY:
This study is an open-label, single ascending dose (SAD) study designed to evaluate the safety and tolerability of ART002g1 in patients with heterozygous familial hypercholesterolemia (HeFH) who require further reduction in low-density lipoprotein cholesterol (LDL-C). ART002g1 uses base editing technology, which is designed to interfere with the expression of the PCSK9 gene in the liver, thereby reducing the circulating levels of PCSK9 and LDL-C. The primary objectives of this study are to determine the safety and pharmacodynamic (PD) profiles of ART002g1 in this patient population.

ELIGIBILITY:
Subjects must meet all the following criteria to be eligible for enrollment:

1. Male or female, aged 18 to 70 years (inclusive) at the time of signing the Informed Consent Form (ICF);
2. Body weight between 45 and 90 kg (inclusive) at screening;
3. Definite diagnosis of heterozygous familial hypercholesterolemia (HeFH), meeting either of the following two criteria (1) or (2):

（1) HeFH diagnosed to be caused by mutations in the LDLR, APOB, or PCSK9 gene;

(2) Meeting 2 out of the 3 following criteria for adults per the Dutch Lipid Clinical Network (DLCN) criteria:

1. Serum LDL-C ≥ 4.7 mmol/L without prior lipid-lowering treatment;
2. Cutaneous or tendinous xanthomas, or arcus cornealis (in subjects < 45 years old);
3. Presence of FH or early-onset atherosclerotic cardiovascular disease (ASCVD) in first-degree relatives.

Subjects must not be enrolled if they meet any one or more of the following exclusion criteria:

1. Diagnosis of compound heterozygous FH, double heterozygous FH, or homozygous FH (HoFH);
2. Positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA titer ≥ 1 × 10² copies/L; positive for hepatitis C virus (HCV) antibody with positive peripheral blood HCV RNA; positive for human immunodeficiency virus (HIV) antibody;
3. Any unstable systemic disease, including but not limited to: unstable angina; cerebrovascular accident or transient ischemic attack (within 6 months prior to screening); myocardial infarction (within 6 months prior to screening); history of heart failure (NYHA Class II-IV); severe arrhythmia requiring pharmacotherapy; liver, kidney, or metabolic diseases; or other unstable systemic diseases as determined by the investigator;
4. History of percutaneous transluminal coronary angioplasty (PTCA), percutaneous coronary intervention (PCI), or coronary artery bypass grafting (CABG) within 6 months prior to the first dose; or documented severe coronary artery stenosis as confirmed by coronary CT or coronary angiography within 90 days prior to randomization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | As of Week 48 (W48) post-administration of ART002g1 for Injection

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Assessments: PK Parameters of ART002g1: Tmax | As of Week 2 (W2) post-administration of ART002g1 for Injection
Pharmacodynamic (PD) Assessments: Serum PCSK9 protein | As of Week 48 (W48) post-administration of ART002g1 for Injection
Pharmacokinetic (PK) Assessments: PK Parameters of ART002g1: Cmax | As of Week 2 (W2) post-administration of ART002g1 for Injection
Pharmacokinetic (PK) Assessments: PK Parameters of ART002g1: AUC | As of Week 2 (W2) post-administration of ART002g1 for Injection
Pharmacokinetic (PK) Assessments: PK Parameters of ART002g1: t½ | As of Week 2 (W2) post-administration of ART002g1 for Injection
Pharmacokinetic (PK) Assessments: PK Parameters of ART002g1: CL | As of Week 2 (W2) post-administration of ART002g1 for Injection
Pharmacokinetic (PK) Assessments: PK Parameters of ART002g1:Vss | As of Week 2 (W2) post-administration of ART002g1 for Injection
Pharmacodynamic (PD) Assessments: Serum LDL-C | As of Week 48 (W48) post-administration of ART002g1 for Injection

CONTACTS AND LOCATIONS:
Overall Officials: Xueying Ding, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Rong Jiang, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No